CLINICAL TRIAL: NCT01398345
Title: Phase 3 Study of Physical Exercise and Respiratory Training as Supportive Treatments for Patients With Severe Chronic Pulmonary Hypertension
Brief Title: Exercise and Respiratory Training as Supportive Treatments for Patients With Chronic Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 364/2003
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Pulmonary Hypertension
MeSH Terms: interventions — Exercise

ARMS (1):
- Exercise and Respiratory Training (Active Comparator)
  Interventions: Behavioral: Exercise and Respiratory Training

INTERVENTIONS:
Behavioral: Exercise and Respiratory Training — Patients in the interventional group will participate in an exercise program 7 days a week at low workloads (10 to 60 W) that will be supervised by physical therapists and physicians.

SUMMARY:
Background

-Pulmonary hypertension (PH) is associated with restricted physical capacity, limited quality of life, and a poor prognosis because of right heart failure. The present study is the first prospective randomized study to evaluate the effects of exercise and respiratory training in patients with severe symptomatic PH.

Methods

-Patients with PH on stable disease-targeted medication will be randomly assigned to a control and a primary training group. Medication will remain unchanged during the study period. Primary end points will be the changes from baseline to week 15 in the distance walked in 6 minutes and in scores of the Short Form Health Survey quality-of-life questionnaire. Changes in WHO functional class, Borg scale, and parameters of echocardiography and gas exchange also will be assessed.

Prospects

-We hope this study will indicate that respiratory and physical training are a promising adjunct to medical treatment in severe PH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe chronic PH who were stable and compensated under optimized medical therapy (such as endothelin antagonists, iloprost, sildenafil, calcium channel blockers, anticoagulants, diuretics, and supplemental oxygen) for at least 3 months before entering the study will be invited to participate.

Additional inclusion criteria will be age of between 18 and 75 years and World Health Organization (WHO) functional class II to IV.

Exclusion Criteria:

* Patients with recent syncope or skeletal or muscle abnormalities prohibiting participation in an exercise program won't be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
distance walked in 6 minutes | baseline - 15 weeks afterwards
change in quality of life as measured by the Short Form Health Survey (SF-36) questionnaire | baseline - 15 weeks afterwards

SECONDARY OUTCOMES:
changes in WHO functional classification | baseline - 15 weeks afterwards
Borg scale assessed immediately after completion of the stress Doppler echocardiography | baseline - 15 weeks afterwards
parameters of echocardiography | baseline - 15 weeks afterwards
parameters of gas exchange | baseline - 15 weeks afterwards

CONTACTS AND LOCATIONS:
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Nagel C, Prange F, Guth S, Herb J, Ehlken N, Fischer C, Reichenberger F, Rosenkranz S, Seyfarth HJ, Mayer E, Halank M, Grunig E. Exercise training improves exercise capacity and quality of life in patients with inoperable or residual chronic thromboembolic pulmonary hypertension. PLoS One. 2012;7(7):e41603. doi: 10.1371/journal.pone.0041603. Epub 2012 Jul 25. PMID 22848542